CLINICAL TRIAL: NCT05974579
Title: A Single Center, Open Label Study to Evaluate Biodistribution, Pharmacokinetics and Safety of [89Zr]Zr-DFO-AP-101 PET (Positron Emission Tomography) in Healthy Volunteers and Amyotrophic Lateral Sclerosis (ALS) Patients
Brief Title: Safety and Dosimetry of a New Radiotracer to Detect Misfolded SOD1 Associated With Amyotrophic Lateral Sclerosis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Collaborators: Eli Lilly and Company (Industry); Chorus Wellness Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-5148; 2024-5148 (Other: CIUSSS de l'Estrie - CHUS)
Record Dates: First submitted 2023-07-11; First posted 2023-08-03 (Actual); Last update posted 2025-01-28 (Actual); Status verified 2025-01

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: PET imaging; CT imaging; AP-101; 89-Zirconium; DFO
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Intervention Model Description: Two groups will be enrolled: 8 healthy subjects and 4 patients with ALS This is non-randomized, all participants will receive the same dose of radiotracer
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy participants (Experimental): Will receive 40MBq of 89Zr-DFO-AP-101, once, at Day 0.
  Interventions: Drug: 89Zr-DFO-AP-101
- Patients with ALS (Experimental): Will receive 40MBq of 89Zr-DFO-AP-101, once, at Day 0.
  Interventions: Drug: 89Zr-DFO-AP-101

INTERVENTIONS:
Drug: 89Zr-DFO-AP-101 — At Day 0, patients will receive one dose of the radiotracer. A PET/CT scan will be done 2h post-dose.
  At 1, 3, 7 and 10 days post-dose, a PET/CT scan will be repeated.

SUMMARY:
Amyotrophic lateral sclerosis (ALS), also known as Lou Gehrig's Disease, is a rare neurodegenerative disease resulting in loss, primarily, of the motor neurons in the motor cortex, brainstem and spinal cord. It currently affects 3 of every 100,000 people in the US.

Currently, there is no diagnostic tool for ALS, resulting in misdiagnosis and significant disease progression before formal diagnosis. An imaging test for early detection of ALS and for monitoring disease progression would have significant diagnostic and prognostic value.

PET imaging with an appropriate radiotracer has great potential as a biomarker for ALS given that it would permit visualization of central nervous system (CNS) pathology in individuals living with the disease.

To that extent, the primary goal of this phase I study is evaluating the safety and biodistribution of the new tracer [89Zr]Zr-DFO-AP-101 in healthy volunteers and ALS patients.

DETAILED DESCRIPTION:
Background: Amyotrophic lateral sclerosis (ALS), also known as Lou Gehrig's Disease, is a rare neurodegenerative disease resulting in loss, primarily, of the motor neurons in the motor cortex, brainstem and spinal cord. It currently affects 3 of every 100,000 people in the US. Currently, there is no diagnostic tool for ALS, resulting in misdiagnosis and significant disease progression before formal diagnosis.

Design: This is a phase I clinical trial and a 2-part, single center, open label study in healthy volunteers (Part A) and confirmed ALS patients (Part B). The primary goal is evaluating the safety and biodistribution of the radiotracer [89Zr]Zr-DFO-AP-101 in healthy volunteers and ALS patients via PET/CT imaging.

Objectives: The primary objectives of this study are:

(Part A) To evaluate, by PET imaging, the safety, biodistribution and dosimetry of [89Zr]Zr-DFO-AP-101 in healthy men and women and in ALS patients

Intervention and Follow-up: Following a screening visit, eligible participants will come to the research center for all study assessments.

* On Day 0, a single intravenous dose of [89Zr]Zr-DFO-AP-101 40 MBq will be administrated and a 45 min whole body PET/CT acquisition will be performed at two hours post injection. Physical exam, ECG, vital signs and blood/urine samples will be collected.
* Further PET acquisitions and same data/samples collection will be repeated at days 1, 3, 7 and 10 post-injection.
* Participants will be contacted for a final follow-up visit approximately 14 days after injection.

ELIGIBILITY:
Inclusion Criteria:

1. Aged of:

   1. For healthy participants: Male or female subjects aged 50 years or older
   2. For ALS patients: Male or female subjects aged 18 years and older
2. Able to remain in a lying position for up to 45 minutes without respiratory support.
3. A) For ALS patients, confirmed diagnostic of definitive ALS according to El-Escorial criteria14 B) for healthy participants: no neurologic condition (confirmed by physical exam)
4. Have venous access sufficient to allow for blood sampling
5. Are reliable and willing to make themselves available for the duration of the study and are willing to follow CRCHUS-specific study procedures.

Exclusion Criteria:

1. Are currently enrolled or were enrolled in the last 12 weeks in any other clinical trial involving a study drug or off label use of a drug or device, or any other type of medical research judged not to be scientifically or medically compatible with this study.
2. Female participants who are pregnant or breast feeding; or women of childbearing potential (<50 years old) and men who are sexually active who are not willing to use an accepted effective contraceptive method.
3. Plan to have surgery or other invasive procedure during the course of the study (up to 14 days post-injection)
4. Have a progressive medical illness including, but not limited to, any cardiovascular, hepatic, respiratory, hematological, endocrine, psychiatric or neurological disease, convulsions, or any clinically significant laboratory abnormality at screening and at first visit (D0) that, in the judgment of the medical doctor, indicate a medical problem that would preclude study participation.
5. Have one of these conditions (for both patient groups):

   1. hepatic disorder such as hepatic encephalopathy, hepatic laboratory abnormalities (ALT or AST ≥3 × ULN or total bilirubin ≥2 × ULN) and hematology abnormalities at screening.
   2. severe chronic kidney disease (eg, an estimated glomerular filtration rate [eGFR] <30 mL/min/1.73m or requires chronic dialysis) at screening.
   3. Have severe active psychiatric illness.
   4. Have a diagnosis of another neurodegenerative disease (e.g. Parkinson disease, Alzheimer's disease, etc).
   5. Have a significant infection or known inflammatory process on screening or at Day 0.
   6. Alcohol or drug abuse based on patient auto-report
   7. Have a history of relevant atopy or drug hypersensitivity or allergy to antibodies;
   8. Have an abnormal blood pressure (supine) defined as a diastolic blood pressure >90 or <45 mmHg and/or a systolic blood pressure >160 or <90 mmHg. Re-testing may occur once during the screening visit within 2 hours of the initial abnormal blood pressure measurement at the discretion of the investigator.
6. For ALS patients:

   1. Have undergone a tracheostomy for ALS symptoms.
   2. Are on nasal intermittent positive pressure ventilation (NIPPV) >4h during the day, while awake for the treatment of ALS related symptoms.
   3. Have other causes of neuromuscular weakness.
7. Have received treatment with biologic agents (such as monoclonal antibodies, including marketed drugs and AP-101) within 3 months or 5 half-lives (whichever is longer) prior to study drug injection.
8. Have received any blood or blood products within the 3 months prior to screening.
9. Cannot communicate reliably with the investigator.
10. Are unwilling or unable to give written informed consent.
11. In the opinion of the medical doctor or his/her delegate, are unsuitable for inclusion in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs) | day 0 (post-injection) to day 14 (end of study)
  Number of adverse events (AEs) and serious adverse events following administration of [89Zr]Zr-DFO-AP-101 that are new or worsened (compared to baseline/pre-dose)
Biodistribution of [89Zr]Zr-DFO-AP-101 | Pre-dose and at 2 hours, 1, 3, 7, 10 days post-dose
  Assessed by whole-body PET imaging
Dosimetry of [89Zr]Zr-DFO-AP-101 in human | Pre-Dose and at 2 hours, 1, 3, 7, 10 days post-dose
  Organ activity concentration (in liver, kidneys, blood, spleen, ...) measured by drawing region of interests on the PET images.

SECONDARY OUTCOMES:
Cmax | Pre-dose and at 2 hours, 1, 3, 7, 10 days post-dose
  Maximal concentration of [89Zr]Zr-DFO-AP-101 in plasma over time after injection
Area under the curve (AUC) | Pre-dose and at 2 hours, 1, 3, 7, 10 days post-dose
  AUC of [89Zr]Zr-DFO-AP-101 in plasma over time after injection
residence time | Pre-dose and at 2 hours, 1, 3, 7, 10 days post-dose
  Time (1/2) of residence of [89Zr]Zr-DFO-AP-101 in plasma
Excretion | Pre-dose and at 2 hours, 1, 3, 7, 10 days post-dose
  Concentration of [89Zr]Zr-DFO-AP-101 urine over time

OTHER OUTCOMES:
Differential labeling and uptake | Pre-dose and at 2 hours, 1, 3, 7, 10 days post-dose
  Assessment of target organ/tissue ratio in ALS patients versus healthy volunteers
differential uptake of neurologic components with the Ultra-High Resolution PET imaging | Pre-dose and at 2hours, 1, 3, 7, 10 dayspost-dose
  SUV values in motor cortex, brainstem and spinal cord, compared between regular PET and UHR PET.

CONTACTS AND LOCATIONS:
Overall Officials: Eric E Turcotte, MD, Study Director — Estrie University Integrated Health and Social Services Center - University Hospital of Sherbrooke; Brigitte Guérin, PhD, Principal Investigator — Estrie University Integrated Health and Social Services Center - University Hospital of Sherbrooke
Locations (1):
- CIUSSS de l'Estrie-CHUS Hospital, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No